CLINICAL TRIAL: NCT00762294
Title: Effect Of Anastrozole And Letrozole On Bone Turnover Markers And Bone Mineral Density In Postmenopausal Women With Primary Breast Cancer: A Pilot Study
Brief Title: Anastrozole and Letrozole
Status: Completed | Type: Observational
Sponsor: UConn Health (Other)
Collaborators: Connecticut Breast Health Initiative (Other)
Responsible Party: Principal Investigator, Pamela Taxel, Associate Professor of Medicine, UConn Health
Other Study IDs: 07-043-2; GCRC # 644
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; arimidex; femara; bone health
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 644-001: Women treated for breast cancer who will be starting Arimidex or Femara

SUMMARY:
Aromatase Inhibitors (AI) are effective for secondary prevention of breast cancer and may soon replace tamoxifen as first-line therapy in the treatment of hormone-sensitive breast cancer. However, because these medications produce a marked reduction in serum estrogen levels, this is likely to result in an increased rate of bone loss and risk of developing osteoporosis and fractures in postmenopausal women treated with these agents. Indeed, substantial bone loss has been reported in several large clinical trials of AIs. Osteoporosis drugs are available that could prevent this loss, but they have frequent side effects and are expensive. Thus, treating all women receiving AIs might not be the most appropriate and cost-effective approach. A better approach might be to select women at highest risk of bone loss and only treat them with antiresorptive agents.

The proposed pilot study will evaluate women who receive anastrozole or letrozole therapy, are receiving adequate amounts of calcium and vitamin D and have baseline normal or moderately low bone mass in order to determine if early changes in bone turnover markers correlate with bone loss at one year. If data from this pilot protocol support our hypothesis, then we would propose a larger trial to confirm it. The ultimate aim is to predict which women are at higher risk of bone loss and therefore treat them earlier with bone-sparing agents, while those with lower risk could be monitored on conservative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with diagnosis of breast cancer - have not started Arimidex or Femara yet, but will be starting .

Exclusion Criteria:

* History of metastasis
* History of chronic kidney
* Liver GI disease
* Disorders affecting calcium metabolism

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women receiving treatment for breast cancer, who will be starting Arimidex or Femara
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2007-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
bone density | baseline, 6 months, 12 months

SECONDARY OUTCOMES:
bone markers | baseline, 1 month, 3 month, 6 month, 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Taxel, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut HEalth Center, Farmington, Connecticut, United States